CLINICAL TRIAL: NCT04977414
Title: A Randomized Controlled Evaluation a Training Intervention to Increase the Use of Statistical Process Control Charts for National Health Service Hospitals in England
Brief Title: Making Data Count Intervention Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Warwick (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Principal Investigator, Kelly Ann Schmidtke, Assistant Professor, University of Warwick
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BSREC 100/20-21
Record Dates: First submitted 2021-07-14; First posted 2021-07-27 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Statistical Process Control Charts

STUDY DESIGN:
Masking Description: Participants cannot be blinded as this is a behavioural intervention.
  Some of the researchers can be blinded. Specifically, it is not possible to blind reviewers R1 and R2 to the board papers group or time-period, as those researchers are extracting charts from the published board papers. R3 and R4 will be blinded and will be instructed to inform R1 if those researchers are unblinded at any point, and whether/how often those researchers are unblinded will be reported in the final manuscript.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist control group (No Intervention): Hospitals assigned to this group will be placed in on a waitlist to receive the training intervention at a later date
- "Making data count" intervention group (Experimental): The Making Data Count training intervention was designed by NHS-Improvement to improve knowledge about SPC charts and to increase their uptake. Training sessions are tailored for two sets of attendees: board members and data analysts. Board member and analyst training sessions are delivered as close as possible in time, typically within the same month. Training sessions for board members are usually delivered over about one-and-a-half hours and focus more heavily on the benefits of control charts compared to other charts. Training sessions for analysts are usually delivered over three hours and focus more heavily on the structure and interpretation of the individual and moving range charts (X-mR charts).
  Interventions: Behavioral: Making Data Count Training intervention

INTERVENTIONS:
Behavioral: Making Data Count Training intervention — The Making Data Count training intervention was designed by NHS-Improvement to improve knowledge about SPC charts and to increase their uptake. Training sessions are tailored for two sets of attendees: board members and data analysts. Board member and analyst training sessions are delivered as close as possible in time, typically within the same month. Training sessions for board members are usually delivered over about one-and-a-half hours and focus more heavily on the benefits of control charts compared to other charts. Training sessions for analysts are usually delivered over three hours and focus more heavily on the structure and interpretation of the individual and moving range charts (X-mR charts).
  Arms: "Making data count" intervention group

SUMMARY:
Hospitals collect copious amounts of data to share with their board for quality assurance and improvement purposes. The way these data are presented can influence board members' decisions. For example, time-series charts highlight the highest and lowest data but do not clarify whether those data lie outside expected or 'common cause' variation. Statistical process control charts make this clarification and, in so doing, guide quality assurance and improvements in a more targeted fashion.

A previous study showed that data suitable for presentation as a control chart are seldom presented in that format. A training intervention called 'Making Data Count' was created to improve the uptake of statistical process control charts by hospitals in England. The current study will use a randomized design to evaluate whether the intervention increases control charts in hospitals that were not early adopters of the training intervention.

This study is a parallel cluster randomized trial (with baseline-line measurements) across 20 National Health Service (NHS) hospitals in England. The hospitals will be randomly split into two groups. One group will be scheduled to experience the training intervention, and the other group will be placed on a waiting list to experience the training later. The primary analysis will compare the difference in the use of control charts between waitlist and intervention hospitals (adjusting for pre-intervention use) reported with 95% confidence intervals. A qualitative thematic analysis of feedback forms will be conducted.

The present research will evaluate the impact of the training intervention on the use of control charts. The results will apply to institutions that are not early adopters of this training intervention.

ELIGIBILITY:
Inclusion Criteria:

* NHS Hospital
* Placed on a red-list for predominantly using R-A-G or two-point data presentations in their board papers.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Gender is not an essential element of this study, as participants randomised I'm the study defined at the level of an NHS Hospital and NHS organisations have no gender or sex.
Enrollment: 15 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in the proportion of SPC charts out of all quality and safety charts from baseline to five months post intervention | One month pre-intervention and then five months post-intervention.
  Change in the proportion of SPC charts (the numerator) out of all charts indicated in each board paper (the denominator)

SECONDARY OUTCOMES:
Chart types | One month pre-intervention and then five months post-intervention.
  counts of whether the charts are time series charts, between subjects charts, time and between charts, or other (e.g., pie)
SPC elements | One month pre-intervention and then five months post-intervention.
  counts of whether the charts include recalculated control lines, highlight special cause variation, use R-A-G colouring, and whether the accesses are labeled.
SPC supporting text | One month pre-intervention and then five months post-intervention.
  counts of whether the charts include recalculated control lines, highlight special counts of whether SPC charts are explained in supporting text, regarding where control lines are set, reasons for variations, and suggestions for improvements.

OTHER OUTCOMES:
Feedback forms | immediately post intervention
  optional forms participants fill out after training to improve future sessions. Intervention group only.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Warwick, Coventry, United Kingdom

REFERENCES:
- [Derived] Schmidtke KA, Kudrna L, Quinn L, Bird P, Hemming K, Venable Z, Lilford R. Cluster randomised evaluation of a training intervention to increase the use of statistical process control charts for hospitals in England: making data count. BMJ Qual Saf. 2025 Aug 18;34(9):621-630. doi: 10.1136/bmjqs-2024-017094. PMID 39237263

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT04977414/Prot_SAP_001.pdf